CLINICAL TRIAL: NCT00366340
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Trial of the Safety, Tolerability, and Immunologic Non-Inferiority of a 13-valent Pneumococcal Conjugate Vaccine Compared to a 7-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in Germany.
Brief Title: Study to Evaluate a 13-valent Pneumococcal Conjugate Vaccine in Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-006
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-06

CONDITIONS: Vaccines, Pneumococcal
Keywords: safety; Vaccine
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- 2 (Active Comparator): 7-valent pneumococcal conjugate vaccine
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — Single 0.5mL dose given at 2, 3, 4 and 11 to 12 months of age
  Arms: 1
Biological: 7-valent pneumococcal conjugate vaccine — Single 0.5mL dose given at 2, 3, 4 and 11 to 12 months of age
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate (13vPnC) vaccine compared to 7-valent pneumococcal conjugate (Prevenar/Prevenar®, 7vPnC), when given concomitantly with Infanrix hexa at 2, 3, 4, months (infant series) and at 11-12 months of age (toddler dose) in Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2 months (56 to 112 days) at time of enrollment.
2. Available for entire study period and whose parent(s) or legal guardian(s) could be reached by telephone.
3. Healthy infant, as determined by medical history, physical examination, and judgment of the investigator.
4. Parent(s) or legal guardian(s) had to be able to complete all relevant study procedures during study participation.

Exclusion criteria:

1. Previous vaccination with licensed or investigational pneumococcal vaccine.
2. Previous vaccination with Hib conjugate, diphtheria, tetanus, pertussis, polio, or hepatitis B vaccines.
3. A previous anaphylactic reaction to any vaccine or vaccine-related component.
4. Contraindication to vaccination with Hib conjugate, diphtheria, tetanus, pertussis, polio, or hepatitis B, or pneumococcal vaccines.
5. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
6. Known or suspected immune deficiency or suppression.
7. History of culture-proven invasive disease caused by S pneumoniae or H influenzae type b.
8. Major known congenital malformation or serious chronic disorder.
9. Significant neurological disorder or history of seizure, including febrile seizure, or significant stable or evolving disorders, such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorders. Did not include resolving syndromes due to birth trauma such as Erb palsy.
10. Receipt of blood products or gamma-globulin (including hepatitis B immunoglobulin and monoclonal antibodies; eg, Synagis®).
11. Participation in another investigational trial. Participation in purely observational studies was acceptable.
12. Infant who was a direct descendant (eg, child or grandchild) of the study site personnel.

Ages: 56 Days to 112 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 604 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com
Locations (44):
- Germany (44):
  - Bad Kreuznach
  - Bad Saulgau
  - Bad Sobernheim
  - Berlin
  - Birkenfeld
  - Bobingen
  - Bramsche
  - Bretten
  - Cham
  - Ehingen
  - Erlangen
  - Eschwege
  - Flensburg
  - Gau-Odernheim
  - Hamburg
  - Herzogenaurach
  - Höchberg
  - Kehl
  - Kiel
  - Kleve
  - Krefeld
  - Ludwigshafen
  - Lübeck
  - Mainz
  - Metzingen
  - Minden
  - Münster
  - NeumÃ¼nster
  - Neumünster
  - Neustadt/Aisch
  - Niebüll
  - Nuremberg
  - Oberkirch
  - Olching
  - Pforzheim
  - Porta Westfalica
  - Ravensburg
  - Tettnang
  - Vellmar
  - Weiden
  - Weilheim
  - Welzheim
  - Wiesbaden
  - Zirndorf

REFERENCES:
- [Derived] Gimenez-Sanchez F, Kieninger DM, Kueper K, Martinon-Torres F, Bernaola E, Diez-Domingo J, Steul K, Juergens C, Gurtman A, Giardina P, Liang JZ, Gruber WC, Emini EA, Scott DA; 501 and 006 study groups. Immunogenicity of a combination vaccine containing diphtheria toxoid, tetanus toxoid, three-component acellular pertussis, hepatitis B, inactivated polio virus, and Haemophilus influenzae type b when given concomitantly with 13-valent pneumococcal conjugate vaccine. Vaccine. 2011 Aug 11;29(35):6042-8. doi: 10.1016/j.vaccine.2011.06.026. Epub 2011 Jun 23. PMID 21704105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Germany from October 2006 to April 2007.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 2, 3, 4 months (infant series) and 12 months of age (toddler dose).
- 7vPnC: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 2, 3, 4 months (infant series) and 12 months of age (toddler dose)
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 301 | 303
Vaccinated Dose 1 | 300 | 303
Vaccinated Dose 2 | 296 | 297
Vaccinated Dose 3 | 294 | 293
Completed | 293 | 293
Not Completed | 8 | 10
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Failure to return | 1 | 0
Period: After the Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 293 | 293
Completed | 290 | 287
Not Completed | 3 | 6
Not completed — Parent/legal guardian request | 1 | 1
Not completed — Failed to return | 0 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 290 | 287
Completed | 289 | 286
Not Completed | 1 | 1
Not completed — Failed to return | 1 | 0
Not completed — Parent/legal guardian request | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 301 | 303 | 604
Age Continuous [Mean (Standard Deviation); unit: months] | 2.5 (0.6) | 2.5 (0.6) | 2.5 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 127 | 278
  Male | 150 | 176 | 326

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥0.35 μg/mL in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series
Description: Percentage of Participants achieving World Health Organization (WHO) predefined antibody threshold ≥0.35 μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after 3-dose infant series (5 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 285 | 279
Percentage of Participants
  Common Serotypes-Serotype 4 | 98.2 [96.0 to 99.4] | 98.2 [95.9 to 99.4]
  Common Serotypes-Serotype 6B | 77.5 [72.2 to 82.2] | 87.1 [82.5 to 90.8]
  Common Serotypes-Serotype 9V | 98.6 [96.4 to 99.6] | 96.4 [93.5 to 98.3]
  Common Serotypes-Serotype 14 | 98.9 [96.9 to 99.8] | 97.5 [94.9 to 99.0]
  Common Serotypes-Serotype 18C | 97.2 [94.5 to 98.8] | 98.6 [96.3 to 99.6]
  Common Serotypes-Serotype 19F | 95.8 [92.7 to 97.8] | 96.0 [93.0 to 98.0]
  Common Serotypes-Serotype 23F | 88.7 [84.5 to 92.2] | 89.5 [85.3 to 92.9]
  Additional Serotypes-Serotype 1 | 96.1 [93.2 to 98.1] | 1.4 [0.4 to 3.7]
  Additional Serotypes-Serotype 3 | 98.2 [95.9 to 99.4] | 6.3 [3.7 to 9.8]
  Additional Serotypes-Serotype 5 | 93.0 [89.3 to 95.6] | 31.6 [25.8 to 37.8]
  Additional Serotypes-Serotype 6A | 91.9 [88.1 to 94.8] | 31.6 [26.1 to 37.5]
  Additional Serotypes-Serotype 7F | 98.6 [96.4 to 99.6] | 4.0 [2.0 to 7.0]
  Additional Serotypes-Serotype 19A | 99.3 [97.5 to 99.9] | 79.2 [73.8 to 83.9]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For serotype 4 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for each common serotype was declared if the lowest limit of the 2-sided 95% CI for the difference between the 2 groups > -10%; Difference = 0.0, 95% CI 2-sided [-2.5 to 2.6]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For serotype 6B the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -9.6, 95% CI 2-sided [-16.0 to -3.3]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For serotype 9V the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 2.2, 95% CI 2-sided [-0.4 to 5.2]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For serotype 14 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 1.5, 95% CI 2-sided [-0.9 to 4.1]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For serotype 18C the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -1.4, 95% CI 2-sided [-4.2 to 1.2]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For serotype 19F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.3, 95% CI 2-sided [-3.8 to 3.3]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For serotype 23F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.8, 95% CI 2-sided [-6.0 to 4.5]

2. Primary Outcome: Geometric Mean Antibody Concentration in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series
Description: Antibody concentration/geometric mean concentration (GMC) as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC ratios (13vPnC/7vPnC) and corresponding 2-sided 95% CI were evaluated.
Time Frame: One month after 3-dose infant series (5 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 285 | 279
μg/mL
  Common Serotypes - Serotype 4 | 2.18 [1.98 to 2.40] | 2.99 [2.68 to 3.33]
  Common Serotypes - Serotype 6B | 0.98 [0.84 to 1.14] | 1.49 [1.27 to 1.75]
  Common Serotypes - Serotype 9V | 1.65 [1.51 to 1.80] | 1.96 [1.77 to 2.17]
  Common Serotypes - Serotype 14 | 4.14 [3.68 to 4.66] | 4.61 [4.07 to 5.23]
  Common Serotypes - Serotype 18C | 1.94 [1.76 to 2.14] | 2.25 [2.04 to 2.49]
  Common Serotypes - Serotype 19F | 1.73 [1.56 to 1.92] | 2.86 [2.53 to 3.24]
  Common Serotypes - Serotype 23F | 1.26 [1.11 to 1.43] | 1.44 [1.25 to 1.65]
  Additional Serotypes - Serotype 1 | 1.83 [1.64 to 2.04] | 0.03 [0.02 to 0.03]
  Additional Serotypes - Serotype 3 | 1.55 [1.41 to 1.72] | 0.05 [0.04 to 0.06]
  Additional Serotypes - Serotype 5 | 1.31 [1.17 to 1.46] | 0.20 [0.18 to 0.23]
  Additional Serotypes - Serotype 6A | 1.33 [1.18 to 1.49] | 0.23 [0.20 to 0.26]
  Additional Serotypes - Serotype 7F | 2.59 [2.36 to 2.85] | 0.04 [0.04 to 0.05]
  Additional Serotypes - Serotype 19A | 3.26 [2.97 to 3.59] | 0.64 [0.58 to 0.71]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For serotype 4 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for each common serotype was declared if the lower limit of the 2-sided 95% CI for the GMC ratio (13vPnC/7vPnC) > 0.5 (2-fold criterion); Ratio = 0.73, 95% CI 2-sided [0.63 to 0.84]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For serotype 6B the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.65, 95% CI 2-sided [0.52 to 0.82]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For serotype 9V the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.84, 95% CI 2-sided [0.74 to 0.96]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For serotype 14 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.90, 95% CI 2-sided [0.76 to 1.07]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For serotype 18C the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 2.25, 95% CI 2-sided [2.04 to 2.49]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For serotype 19F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.60, 95% CI 2-sided [0.51 to 0.71]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For serotype 23F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio = 0.88, 95% CI 2-sided [0.73 to 1.06]

3. Primary Outcome: Percentage of Participants Achieving Antibody Titer ≥1:8 as Measured by Opsonophagocytic Activity Assay (OPA) in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series.
Description: Percentage of Participants achieving functional antibody titer ≥1:8 as measured by opsonophagocytic activity assay (OPA) along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after 3-dose infant series (5 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n)=number of participants with a determinate postinfant series OPA antibody titer to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 285 | 279
Percentage of Participants
  Common Serotypes - Serotype 4 (n=92,94) | 100.0 [96.1 to 100.0] | 100.0 [96.2 to 100.0]
  Common Serotypes - Serotype 6B (n=100,94) | 96.0 [90.1 to 98.9] | 98.9 [94.2 to 100.0]
  Common Serotypes - Serotype 9V (n=89,89) | 100.0 [95.9 to 100.0] | 100.0 [95.9 to 100.0]
  Common Serotypes - Serotype 14 (n=95,89) | 100.0 [96.2 to 100.0] | 100.0 [95.9 to 100.0]
  Common Serotypes - Serotype 18C (n=100,94) | 100.0 [96.4 to 100.0] | 98.9 [94.2 to 100.0]
  Common Serotypes - Serotype 19F (n=100,94) | 96.0 [90.1 to 98.9] | 93.6 [86.6 to 97.6]
  Common Serotypes - Serotype 23F (n=100,93) | 96.0 [90.1 to 98.9] | 95.7 [89.4 to 98.8]
  Additional Serotypes - Serotype 1 (n=100,92) | 93.0 [86.1 to 97.1] | 4.3 [1.2 to 10.8]
  Additional Serotypes - Serotype 3 (n=100,94) | 99.0 [94.6 to 100.0] | 24.5 [16.2 to 34.4]
  Additional Serotypes - Serotype 5 (n=100,94) | 99.0 [94.6 to 100.0] | 4.3 [1.2 to 10.5]
  Additional Serotypes - Serotype 6A (n=99,93) | 96.0 [90.0 to 98.9] | 72.0 [61.8 to 80.9]
  Additional Serotypes - Serotype 7F (n=99,94) | 100.0 [96.3 to 100.0] | 78.7 [69.1 to 86.5]
  Additional Serotypes - Serotype 19A (n=95,94) | 100.00 [96.2 to 100.0] | 17.0 [10.1 to 26.2]

4. Primary Outcome: Geometric Mean Antibody Titer in 13vPnC Group Relative to 7vPnC Group After the 3-Dose Infant Series
Description: Antibody functionality/geometric mean titer (GMT) as measured by opsonophagocytic activity assay (OPA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after 3-dose infant series (5 months of age)
Population: Evaluable immunogenicity (per protocol) population of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n)= number of participants with a determinate antibody titer for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 285 | 279
titer
  Common Serotypes -Serotype 4 (n=92,94) | 1573.29 [1283.03 to 1929.21] | 1860.79 [1540.00 to 2248.41]
  Common Serotypes - Serotype 6B (n=100,94) | 744.43 [556.91 to 995.11] | 1160.76 [921.46 to 1462.19]
  Common Serotypes - Serotype 9V (n=89,89) | 4937.84 [3614.78 to 6745.14] | 5379.51 [3935.51 to 7353.34]
  Common Serotypes - Serotype 14 (n=95,89) | 2139.65 [1570.10 to 2915.79] | 3345.19 [2473.27 to 4524.50]
  Common Serotypes - Serotype 18C (n=100,94) | 1509.65 [1243.64 to 1832.56] | 1780.26 [1382.42 to 2292.59]
  Common Serotypes - Serotype 19F (n=100,94) | 150.12 [116.89 to 192.81] | 165.69 [122.98 to 223.23]
  Common Serotypes - Serotype 23F (n=100,93) | 1089.92 [795.20 to 1493.86] | 1070.83 [786.59 to 1457.78]
  Additional Serotypes - Serotype 1 (n=100,92) | 50.21 [39.39 to 64.02] | 4.15 [3.99 to 4.32]
  Additional Serotypes - Serotype 3 (n=100,94) | 250.73 [205.52 to 305.89] | 6.13 [5.17 to 7.28]
  Additional Serotypes - Serotype 5 (n=100,94) | 162.02 [126.31 to 207.82] | 4.64 [3.96 to 5.43]
  Additional Serotypes - Serotype 6A (n=99,93) | 1228.45 [883.49 to 1708.11] | 122.40 [74.09 to 202.21]
  Additional Serotypes - Serotype 7F (n=99,94) | 11544.75 [9364.02 to 14233.34] | 115.45 [75.16 to 177.32]
  Additional Serotypes - Serotype 19A (n=95,94) | 442.48 [360.53 to 543.06] | 6.70 [5.19 to 8.66]

5. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Haemophilus Influenzae Type b, Diphtheria Toxoid, and Hepatitis B in 13vPnC Group Relative to 7vPnC Group After the Infant Series and After the Toddler Dose
Description: Predefined Antibody Levels for Haemophilus Influenzae Type b (0.15 µg/mL or 1.0 µg/mL), for Diphtheria Toxoid (0.01 or 0.1 International units [IU]/mL) and for Hepatitis B (≥ 10.0 mIU/mL).
Time Frame: One month after the infant series (5 months of age) ; one month after the toddler dose (13 months of age)
Population: Evaluable immunogenicity (per protocol) population of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (N)= number of participants with a antibody concentration ≥ the prespecified level for the given concomitant antigen.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- 13vPnC After Infant Series: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 2, 3, 4 months (infant series).
- 7vPnC After Infant Series: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 2, 3, 4 months (infant series).
- 13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 12 months of age (toddler dose).
- 7vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 12 months of age (toddler dose)
Arm/Group | 13vPnC After Infant Series | 7vPnC After Infant Series | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 267 | 252 | 252 | 242
Percentage of Participants
  Haemophilus influenzae type b 0.15 µg/mL threshold | 89.5 [85.2 to 92.9] | 86.9 [82.1 to 90.8] | 100.0 [98.5 to 100.0] | 100.0 [98.5 to 100.0]
  Haemophilus influenzae type b 1.0 µg/mL threshold | 58.4 [52.3 to 64.4] | 54.0 [47.6 to 60.2] | 99.6 [97.8 to 100.0] | 97.9 [95.2 to 99.3]
  Diphtheria toxoid at 0.01 IU/mL threshold | 100.0 [98.7 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0]
  Diphtheria toxoid at 0.1 IU/mL threshold | 89.7 [85.5 to 93.0] | 94.2 [90.6 to 96.7] | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0]
  Hepatitis B at ≥ 10.0 mIU/mL | 94.9 [91.7 to 97.2] | 96.3 [93.2 to 98.2] | 99.3 [97.4 to 99.9] | 98.5 [96.1 to 99.6]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.15 µg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) > -10%; Difference = 2.6, 95% CI 2-sided [-3.0 to 8.3]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Haemophilus influenzae type b the difference in percentages between the two groups (13vPnC - 7vPnC) at 1.0 µg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 4.5, 95% CI 2-sided [-4.1 to 13.0]
Statistical Analysis 3: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For diphtheria toxoid the difference in percentages between the two groups(13vPnC - 7vPnC) at 0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.0, 95% CI [-1.4 to 1.5]
Statistical Analysis 4: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For diphtheria toxoid the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.1 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -4.5, 95% CI [-9.3 to 0.3]
Statistical Analysis 5: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Haemophilus Influenzae Type b the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.15 µg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.0, 95% CI 2-sided [-1.5 to 1.5]
Statistical Analysis 6: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For hepatitis B the difference in percentages between the two groups (13vPnC - 7vPnC) at ≥ 10.0 mIU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -1.3, 95% CI [-5.0 to 2.3]
Statistical Analysis 7: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 5, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 1.7, 95% CI 2-sided [-0.4 to 4.4]
Statistical Analysis 8: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For diphtheria toxoid the difference in percentages between the two groups (13vPnC - 7vPnC) at 0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 9: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 5, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 10: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; [analysis description as in outcome 5, analysis 6]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.8, 95% CI [-1.3 to 3.3]

6. Primary Outcome: Geometric Mean Antibody Concentration of Haemophilus Influenzae Type b in 13vPnC Group Relative to 7vPnC Group After the Infant Series and After the Toddler Dose
Time Frame: One month after the infant series (5 months of age) ; one month after the toddler dose (13 months of age)
Population: Evaluable immunogenicity (per protocol) population of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (N)= number of participants with a determinate antibody concentration for the specified concomitant antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- 13vPnC AfterToddler Dose: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 12 months of age (toddler dose).
- 7vPnC AfterToddler Dose: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 12 months of age (toddler dose)
Arm/Group | 13vPnC After Infant Series | 7vPnC After Infant Series | 13vPnC AfterToddler Dose | 7vPnC AfterToddler Dose
Number analyzed (Participants) | 267 | 252 | 285 | 279
μg/mL | 1.23 [1.03 to 1.46] | 1.00 [0.83 to 1.20] | 11.79 [10.36 to 13.41] | 10.24 [8.88 to 11.82]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Haemophilus influenzae type b the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for the concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the GMC ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 1.23, 95% CI 2-sided [0.96 to 1.58]
Statistical Analysis 2: Comparison: 13vPnC AfterToddler Dose vs 7vPnC AfterToddler Dose; For Haemophilus influenzae type b µg/mL the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 1.15, 95% CI 2-sided [0.95 to 1.39]

7. Primary Outcome: Geometric Mean Antibody Concentration of Diphtheria Toxoid in 13vPnC Group Relative to 7vPnC Group After the Infant Series and After the Toddler Dose
Time Frame: One month after the infant series (5 months of age) ; one month after the toddler dose (13 months of age)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC After Infant Series | 7vPnC After Infant Series | 13vPnC AfterToddler Dose | 7vPnC AfterToddler Dose
Number analyzed (Participants) | 272 | 258 | 285 | 279
IU/mL | 0.36 [0.32 to 0.41] | 0.53 [0.47 to 0.60] | 2.67 [2.44 to 2.93] | 3.08 [2.74 to 3.47]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For diphtheria toxoid the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.68, 95% CI 2-sided [0.57 to 0.80]
Statistical Analysis 2: Comparison: 13vPnC AfterToddler Dose vs 7vPnC AfterToddler Dose; For diphtheria toxoid the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.87, 95% CI 2-sided [0.75 to 1.01]

8. Primary Outcome: Geometric Mean Antibody Concentration of Hepatitis B in 13vPnC Group Relative to 7vPnC Group After the Infant Series and After the Toddler Dose
Description: Antibody geometric mean concentration (GMC) as measured by mcg/mL for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after the infant series (5 months of age) ; one month after the toddler dose (13 months of age)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 13vPnC After Infant Series | 7vPnC After Infant Series | 13vPnC AfterToddler Dose | 7vPnC AfterToddler Dose
Number analyzed (Participants) | 277 | 268 | 285 | 279
mIU/mL | 145.19 [122.62 to 171.92] | 165.25 [140.33 to 194.61] | 1118.05 [935.26 to 1336.56] | 1195.82 [976.12 to 1464.98]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For hepatitis B the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.88, 95% CI 2-sided [0.69 to 1.11]
Statistical Analysis 2: Comparison: 13vPnC AfterToddler Dose vs 7vPnC AfterToddler Dose; For hepatitis B the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Ratio = 0.93, 95% CI 2-sided [0.71 to 1.22]

9. Primary Outcome: Geometric Mean Concentration in 13vPnC Group Relative to 7vPnC Group Before and After the Toddler Dose
Description: Antibody concentration/geometric mean concentration as measured by ELISA with their corresponding 95% CI immediately before and after the toddler dose for 7 common pneumococcal serotypes (Serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: Immediately before (12 months of age) and one month after the toddler dose (13 months of age)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- 13vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 2, 3, 4 months (infant series).
- 7vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 2, 3, 4 months (infant series).
Arm/Group | 13vPnC Before Toddler Dose | 7vPnC Before Toddler Dose | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 285 | 279 | 285 | 279
μg/mL
  Common Serotypes -Serotype 4 (n=277,264,276,263) | 0.46 [0.42 to 0.51] | 0.58 [0.53 to 0.64] | 4.16 [3.75 to 4.62] | 5.07 [4.53 to 5.67]
  Common Serotypes - Serotype 6B (n=275,261,273,251) | 0.97 [0.87 to 1.07] | 1.06 [0.94 to 1.20] | 9.14 [8.14 to 10.26] | 9.85 [8.66 to 11.22]
  Common Serotypes - Serotype 9V (n=277,265,277,262) | 0.46 [0.42 to 0.50] | 0.52 [0.48 to 0.57] | 2.75 [2.52 to 2.99] | 3.36 [3.02 to 3.73]
  Common Serotypes - Serotype 14 (n=273,263,276,260) | 2.20 [1.96 to 2.48] | 2.65 [2.34 to 3.00] | 8.34 [7.50 to 9.28] | 11.01 [9.87 to 12.29]
  Common Serotypes-Serotype 18C (n=277,265,276,263) | 0.33 [0.30 to 0.36] | 0.39 [0.36 to 0.43] | 2.79 [2.53 to 3.07] | 3.44 [3.08 to 3.84]
  Common Serotypes-Serotype 19F (n=276,264,276,263) | 0.68 [0.60 to 0.76] | 0.58 [0.52 to 0.66] | 5.99 [5.36 to 6.68] | 4.72 [4.12 to 5.41]
  Common Serotypes-Serotype 23F (n=275,264,277,264) | 0.33 [0.30 to 0.37] | 0.39 [0.34 to 0.45] | 3.36 [2.98 to 3.78] | 4.33 [3.75 to 5.00]
  Additional - Serotype 1 (n=277,264,278,257) | 0.52 [0.48 to 0.57] | 0.03 [0.02 to 0.03] | 4.25 [3.80 to 4.75] | 0.03 [0.03 to 0.04]
  Additional - Serotype 3 (n=275,264,278,255) | 0.25 [0.23 to 0.28] | 0.05 [0.05 to 0.06] | 1.02 [0.92 to 1.13] | 0.07 [0.06 to 0.08]
  Additional - Serotype 5 (n=275,264,276,220) | 0.74 [0.67 to 0.81] | 0.34 [0.30 to 0.39] | 3.56 [3.25 to 3.89] | 0.51 [0.45 to 0.58]
  Additional - Serotype 6A (n=276,264,274,255) | 0.76 [0.68 to 0.85] | 0.33 [0.29 to 0.37] | 5.88 [5.24 to 6.59] | 1.74 [1.51 to 2.01]
  Additional - Serotype 7F (n=277,264,278,263) | 0.99 [0.91 to 1.08] | 0.04 [0.04 to 0.04] | 4.79 [4.29 to 5.34] | 0.05 [0.04 to 0.05]
  Additional - Serotype 19A (n=277,264,271,260) | 1.28 [1.14 to 1.45] | 0.72 [0.65 to 0.80] | 9.58 [8.68 to 10.58] | 3.79 [3.40 to 4.21]

10. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (Sig) (present and interfered with limb movement). Induration and erythema were scaled as Any (induration or erythema present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (Mod)(2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Day 1 through 4 after each dose
Population: Safety population, included participants who received given dose; (n) = number of participants reporting the specific characteristic.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 2 months (infant series).
- 7vPnC Dose 1: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 2 months (infant series).
- 13vPnC Dose 2: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 3 months (infant series).
- 7vPnC Dose 2: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 3 months (infant series).
- 13vPnC Dose 3: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 4 months (infant series).
- 7vPnC Dose 3: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 4 months (infant series).
- 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 12 months of age.
- 7vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with combined Diphtheria-Tetanus-acellular Pertussis (DTPa), Hepatitis B, Poliovirus and Haemophilus influenzae type b vaccine (Infanrix hexa) at 12 months of age.
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 300 | 303 | 296 | 297 | 294 | 293 | 290 | 287
percentage of participants
  Tenderness-Any (n=267,267,250,241,229,221,206,96) | 33.0 | 32.6 | 29.2 | 31.5 | 27.1 | 21.3 | 53.4 | 51.9
  Tenderness-Sig (n=260,258,236,226,215,209,176,158) | 7.7 | 7.0 | 4.7 | 7.5 | 4.2 | 2.9 | 10.8 | 12.7
  Swelling-Any (n=266,263,244,242,226,224,190,176) | 28.2 | 20.5 | 26.6 | 35.1 | 26.1 | 28.6 | 36.8 | 43.8
  Swelling-Mild (n=265,263,243,239,226,223,186,172) | 24.5 | 19.0 | 24.3 | 33.5 | 24.8 | 27.8 | 33.3 | 40.7
  Swelling-Mod (n=261,256,235,227,217,211,174,158) | 7.3 | 5.9 | 7.7 | 6.6 | 6.9 | 5.2 | 12.1 | 12.7
  Swelling-Severe(n=259,255,232,223,214,208,166,152) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Redness-Any (n=266,272,247,252,238,231,196,184) | 28.2 | 36.4 | 34.4 | 46.8 | 34.9 | 39.8 | 47.4 | 56.0
  Redness-Mild (n=265,271,247,250,237,229,191,180) | 27.2 | 36.2 | 33.6 | 45.6 | 34.2 | 38.9 | 44.5 | 52.8
  Redness-Mod (n=260,256,232,224,217,210,173,158) | 1.9 | 1.6 | 1.7 | 3.6 | 4.6 | 2.4 | 11.6 | 15.2
  Redness-Severe (n=259,255,232,222,214,208,166,153) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.7

11. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events (Infant Series)
Description: Systemic events (any fever ≥ 38 degrees Celsius [C], decreased appetite, irritability, increased sleep, decreased sleep, and hives [urticaria]) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Day 1 through 4 after each dose
Population: Safety population, participants who received given dose; (n)= number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3
Number analyzed (Participants) | 300 | 303 | 296 | 297 | 294 | 293
percentage of participants
  Fever ≥38°C but ≤ 39°C (n=269,266,248,250,242,232) | 43.5 | 38.7 | 46.8 | 48.4 | 46.3 | 36.6
  Fever >39°C but ≤40°C (n=260,256,238,225,216,210) | 4.2 | 1.6 | 8.8 | 4.4 | 3.7 | 1.4
  Fever >40°C (n=259,256,233,223,216,209) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Decreased Appetite (n=269,267,249,245,236,225) | 33.1 | 30.3 | 33.7 | 34.3 | 33.1 | 30.2
  Irritability (n=275,266,254,252,238,235) | 42.5 | 45.1 | 47.2 | 55.2 | 45.4 | 48.9
  Increased Sleep (n=284,272,258,256,240,241) | 61.6 | 58.8 | 53.9 | 66.8 | 49.6 | 49.4
  Decreased Sleep (n=266,264,240,234,230,221) | 25.2 | 26.1 | 23.8 | 23.1 | 20.9 | 24.4
  Meds to Prevent Sx (n=261,262,237,234,220,220) | 8.8 | 9.5 | 10.1 | 15.4 | 10.0 | 15.0
  Meds to Treat Sx (n=263,266,244,235,226,225) | 20.2 | 21.1 | 28.3 | 27.2 | 20.8 | 19.1

12. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events (Toddler Series)
Description: as for outcome 11
Time Frame: Day 1 through 4 after each dose
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 290 | 287
percentage of participants
  Fever ≥38°C but ≤ 39°C (n=206,200) | 58.7 | 62.0
  Fever >39°C but ≤40°C (n=174,157) | 12.6 | 8.9
  Fever >40°C (n=166,152) | 0.6 | 0.0
  Decreased Appetite (n=204,192) | 43.6 | 46.4
  Irritability (n=213,200) | 55.4 | 61.0
  Increased Sleep (n=202,197) | 56.4 | 54.8
  Decreased Sleep (n=195,170) | 31.8 | 28.8
  Medication to Prevent Symptoms (n=184,182) | 32.1 | 33.0
  Medication to Treat Symptoms (n=178,167) | 18.0 | 18.6

ADVERSE EVENTS:
Groups:
- 13vPnC Infant Series: Participants received one single 0.5mL dose of 13vPnC coadministered with Infanrix hexa at 2, 3, 4 months. Adverse events were collected from dose 1 to approximately one month after dose 3.
- 7vPnC Infant Series: Participants received one single 0.5mL dose of 7vPnC coadministered with Infanrix hexa at 2, 3, 4 months. Adverse events were collected from dose 1 to approximately one month after dose 3.
- 13vPnC Post-Infant Series: Participants received one single 0.5mL dose of 13vPnC coadministered with Infanrix hexa at 2, 3, 4 months. Adverse events were collected from approximately one month after dose 3 to toddler dose.
- 7vPnC Post-Infant Series: Participants received one single 0.5mL dose of 7vPnC coadministered with Infanrix hexa at 2, 3, 4 months (infant series) and 12 months of age (toddler dose). Adverse events were collected from approximately one month after dose 3 to toddler dose.
- 13vPnC Toddler Dose: Participants received one single 0.5mL dose of 13vPnC at 12 months of age. Adverse events were collected for approximately one month after toddler dose.
- 7vPnC Toddler Dose: Participants received one single 0.5mL dose of 7vPnC coadministered with Infanrix hexa at 12 months of age. Adverse events were collected for approximately one month after toddler dose.
- 13vPnC 6-Month Follow-up: Participants received one single 0.5mL dose of 13vPnC coadministered with Infanrix hexa at 2, 3, 4 months (infant series) and 12 months of age (toddler dose). Adverse events were collected for approximately six months after last visit.
- 7vPnC 6-Month Follow-up: Participants received one single 0.5mL dose of 7vPnC coadministered with Infanrix hexa at 2, 3, 4 months (infant series) and 12 months of age (toddler dose). Adverse events were collected for approximately six months after last visit.
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC Post-Infant Series | 7vPnC Post-Infant Series | 13vPnC Toddler Dose | 7vPnC Toddler Dose | 13vPnC 6-Month Follow-up | 7vPnC 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 12/300 | 10/303 | 21/300 | 23/303 | 3/300 | 4/303 | 11/300 | 14/303
Other Adverse Events (participants affected / at risk) | 220/299 | 225/300 | 13/299 | 25/300 | 152/289 | 143/284 | 11/287 | 8/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=300) | 7vPnC Infant Series (N=303) | 13vPnC Post-Infant Series (N=300) | 7vPnC Post-Infant Series (N=303) | 13vPnC Toddler Dose (N=300) | 7vPnC Toddler Dose (N=303) | 13vPnC 6-Month Follow-up (N=300) | 7vPnC 6-Month Follow-up (N=303)
Accidental exposure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 4 | 1 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 4 | 1 | 1 | 3 | 3
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 2 | 2 | 2 | 3 | 1 | 1 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nicotine poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Viral tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=299) | 7vPnC Infant Series (N=300) | 13vPnC Post-Infant Series (N=299) | 7vPnC Post-Infant Series (N=300) | 13vPnC Toddler Dose (N=289) | 7vPnC Toddler Dose (N=284) | 13vPnC 6-Month Follow-up (N=287) | 7vPnC 6-Month Follow-up (N=287)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Congenital torticollis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Craniotabes (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hereditary fructose intolerance (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Macrocephaly (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Naevus flammeus (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear disorder (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Otosalpingitis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 22 | 25 | 0 | 0 | 9 | 6 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pupils unequal (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryoadenitis acquired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 14 | 0 | 0 | 4 | 8 | 1 | 0
Flatulence (Gastrointestinal disorders) | 11 | 8 | 0 | 0 | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 11 | 6 | 0 | 0 | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 7 | 0 | 0 | 3 | 2 | 0 | 0
Teething (Gastrointestinal disorders) | 6 | 8 | 0 | 2 | 4 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Anal prolapse (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 29 | 27 | 0 | 0 | 14 | 28 | 0 | 0
Injection site swelling (General disorders) | 3 | 4 | 0 | 0 | 3 | 5 | 0 | 0
Injection site erythema (General disorders) | 2 | 2 | 0 | 0 | 4 | 5 | 0 | 0
Injection site induration (General disorders) | 1 | 3 | 0 | 0 | 1 | 4 | 0 | 0
Injection site pain (General disorders) | 1 | 1 | 0 | 0 | 2 | 4 | 0 | 0
Injection site reaction (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 75 | 64 | 2 | 1 | 40 | 32 | 0 | 0
Bronchitis (Infections and infestations) | 49 | 45 | 2 | 2 | 20 | 19 | 0 | 0
Rhinitis (Infections and infestations) | 24 | 32 | 2 | 0 | 16 | 13 | 0 | 0
Nasopharyngitis (Infections and infestations) | 19 | 28 | 0 | 1 | 10 | 14 | 0 | 0
Gastroenteritis (Infections and infestations) | 21 | 22 | 0 | 0 | 16 | 11 | 0 | 0
Viral infection (Infections and infestations) | 11 | 14 | 0 | 0 | 5 | 8 | 0 | 0
Oral candidiasis (Infections and infestations) | 9 | 12 | 0 | 1 | 1 | 3 | 0 | 0
Otitis media (Infections and infestations) | 7 | 13 | 0 | 0 | 12 | 10 | 0 | 0
Febrile infection (Infections and infestations) | 7 | 10 | 0 | 1 | 7 | 5 | 0 | 0
Candida nappy rash (Infections and infestations) | 4 | 5 | 0 | 1 | 2 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 6 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 3 | 5 | 0 | 0 | 1 | 1 | 0 | 0
Exanthema subitum (Infections and infestations) | 4 | 4 | 0 | 0 | 3 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 4 | 0 | 0 | 1 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 3 | 0 | 0
Skin candida (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Varicella (Infections and infestations) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Viral rash (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Eczema infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudocroup (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Scarlet fever (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinobronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0
Feeding disorder neonatal (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia neonatal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Coordination abnormal (Nervous system disorders) | 3 | 7 | 0 | 1 | 0 | 2 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertonia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 1
High-pitched crying (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Myotonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crying (Psychiatric disorders) | 11 | 10 | 0 | 0 | 1 | 2 | 0 | 0
Restlessness (Psychiatric disorders) | 7 | 14 | 0 | 0 | 3 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 3 | 3 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 5 | 7 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 0 | 0 | 7 | 3 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraclavicular retraction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 22 | 25 | 0 | 1 | 17 | 16 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 10 | 14 | 2 | 0 | 3 | 5 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 6 | 6 | 1 | 0 | 3 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 7 | 5 | 0 | 2 | 3 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 0 | 0 | 1 | 3 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 0 | 2 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 3 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mastocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atopy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Granuloma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Omphalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinolaryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Accidental exposure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fine motor delay (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudoparalysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Screaming (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
21-hydroxylase deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood immunoglobulin e increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Developmental delay (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 88/267 | 87/267 | 0/0 | 0/0 | 110/206 | 96/185 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (Any)
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 73/250 | 76/241 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (Any)
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 62/229 | 47/221 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (Any)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 20/260 | 18/258 | 0/0 | 0/0 | 19/176 | 20/158 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (Significant)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 11/236 | 17/226 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (Significant)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 9/215 | 6/209 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (Significant)
Induration (Any) (Skin and subcutaneous tissue disorders) | 75/266 | 54/263 | 0/0 | 0/0 | 70/190 | 77/176 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (Any)
Induration (Any) (Skin and subcutaneous tissue disorders) | 65/244 | 85/242 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (Any)
Induration (Any) (Skin and subcutaneous tissue disorders) | 59/226 | 64/224 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (Any)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 65/265 | 50/263 | 0/0 | 0/0 | 62/186 | 70/172 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (Mild)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 59/243 | 80/239 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (Mild)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 56/226 | 62/223 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (Mild)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 19/261 | 15/256 | 0/0 | 0/0 | 21/174 | 20/158 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (Moderate)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 18/235 | 15/227 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (Moderate)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 15/217 | 11/211 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (Moderate)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/259 | 0/255 | 0/0 | 0/0 | 0/166 | 0/152 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (Severe)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/232 | 0/223 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (Severe)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/214 | 0/208 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (Severe)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 75/266 | 99/272 | 0/0 | 0/0 | 93/196 | 103/184 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (Any)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 85/247 | 118/252 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (Any)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 83/238 | 92/231 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Any)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 72/265 | 98/271 | 0/0 | 0/0 | 85/191 | 95/180 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (Mild)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 83/247 | 114/250 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (Mild)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 81/237 | 89/229 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Mild)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 5/260 | 4/256 | 0/0 | 0/0 | 20/173 | 24/158 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (Moderate)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 4/232 | 8/224 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (Moderate)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 10/217 | 5/210 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Moderate)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/259 | 0/255 | 0/0 | 0/0 | 0/166 | 1/153 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (Severe)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/232 | 0/222 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (Severe)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/214 | 0/208 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Severe)
Fever ≥38°C but ≤39°C (General disorders) | 117/269 | 103/266 | 0/0 | 0/0 | 121/206 | 124/200 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 116/248 | 121/250 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 112/242 | 85/232 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38°C but ≤39°C
Fever >39°C but ≤40°C (General disorders) | 11/260 | 4/256 | 0/0 | 0/0 | 22/174 | 14/157 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 21/238 | 10/225 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 8/216 | 3/210 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39°C but ≤40°C
Fever >40°C (General disorders) | 0/259 | 0/256 | 0/0 | 0/0 | 1/166 | 0/152 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40°C
Fever >40°C (General disorders) | 0/233 | 0/223 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40°C
Fever >40°C (General disorders) | 2/216 | 0/209 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40°C
Decreased appetite (General disorders) | 89/269 | 81/267 | 0/0 | 0/0 | 89/204 | 89/192 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 84/249 | 84/245 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 78/236 | 68/225 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 117/275 | 120/266 | 0/0 | 0/0 | 118/213 | 122/200 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 120/254 | 139/252 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 108/238 | 115/235 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 175/284 | 160/272 | 0/0 | 0/0 | 114/202 | 108/197 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 139/258 | 171/256 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 119/240 | 119/241 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 67/266 | 69/264 | 0/0 | 0/0 | 62/195 | 49/170 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 57/240 | 54/234 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 48/230 | 54/221 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.